CLINICAL TRIAL: NCT00354952
Title: Impact of Azithromycin and Clarithromycin Therapy on Pharyngeal Carriage of Macrolide-Resistant Streptococci Among Healthy Volunteers: A Randomised, Double-Blind, Placebo-Controlled Trial
Brief Title: Selection of Antibiotic Resistance by Azithromycin and Clarithromycin in the Oral Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: UA-Med Micro-2002
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2003-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Antibiotic exposure; Resistance selection
MeSH Terms: interventions — Macrolides; Azithromycin; Clarithromycin

INTERVENTIONS:
Drug: Macrolides (azithromycin or clarithromycin)

SUMMARY:
Resistance to antibiotics is a major public-health problem and studies linking antibiotic use and resistance have shown an association not a causal effect. Utilizing the newer macrolides, azithromycin and clarithromycin that are commonly prescribed for respiratory infections, we investigated the direct impact of antibiotic exposure on resistance at the individual level.

DETAILED DESCRIPTION:
Resistance to antibiotics is a major public-health problem and studies linking antibiotic use and resistance have shown an association not a causal effect. Utilizing the newer macrolides, azithromycin and clarithromycin that are commonly prescribed for respiratory infections, we investigated the direct impact of antibiotic exposure on resistance at the individual level. 203 healthy cohorts were treated with azithromycin, clarithromycin, or a placebo in a randomised, double-blind trial. Pharyngeal swabs were collected pre- (day 0) and post-antibiotic administration (days 8, 14, 28, 42, 180) and proportions of macrolide-resistant streptococci (MRS) were determined at each time-point.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults (≥ 18 years of age)
* non-pregnant
* free of any respiratory tract infection
* not having been administered any antibiotic at least in the past three months

Exclusion Criteria:

* <18 years of age
* pregnant
* having a respiratory tract infection
* having been administered any antibiotic at least in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203
Dates: Start 2002-07; Study Completion 2003-10

PRIMARY OUTCOMES:
Changes in proportions of macrolide-resistant streptococcal (MRS) carriage in the oropharynx

SECONDARY OUTCOMES:
Variations in the carriage of macrolide-resistance genes due to macrolide exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Goossens, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Depatment of Medical Microbiology, Universiteit Antwerpen, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Malhotra-Kumar S, Lammens C, Coenen S, Van Herck K, Goossens H. Effect of azithromycin and clarithromycin therapy on pharyngeal carriage of macrolide-resistant streptococci in healthy volunteers: a randomised, double-blind, placebo-controlled study. Lancet. 2007 Feb 10;369(9560):482-90. doi: 10.1016/S0140-6736(07)60235-9. PMID 17292768